CLINICAL TRIAL: NCT06638424
Title: Study of the Impact of Cataract Surgery on the Corneal Epithelium and Ocular Surface of Diabetic Patients
Acronym: CATARA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9246
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cataract Diabetic
Keywords: Cataract; Diabetes; Corneal epithelium; Lacrimal gland; Corneal neuropathy; Meibomian dysfunction
MeSH Terms: conditions — Cataract; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetes is one of the most common fatal metabolic diseases in the world. Diabetes-induced ocular surface alterations are poorly understood. Indeed, it was once thought that the cornea, avascular, was immune to the effects of diabetes. A growing number of publications now demonstrate the opposite. These alterations affect up to 70% of diabetic patients at some point in the progression of their diabetes.

Another common complication of diabetes is the early development of a cataract, requiring surgery. Diabetic patients are therefore more likely to require surgery at an early age than the general population.

Diabetes and cataract surgery both induce corneal changes. Cataract surgery in diabetic patients is therefore at greater risk of corneal complications. Diabetes induces dysfunction of the main lacrimal gland, corneal neuropathy, meibomian dysfunction and a decrease in conjunctival mucus cells. Diabetic patients are therefore particularly at risk of exacerbation or appearance of alterations of the corneal epithelium and the ocular surface in postoperative cataract surgery.

Therefore, it seems necessary to evaluate the impact of cataract surgery on the ocular surface and corneal epithelium of diabetic patients, in order to improve their management.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years);
* Patient operated on for cataract at HUS between January 2022 and January 2024;
* Patient who did not express his opposition to the reuse of his data for scientific research purposes;
* Patient who benefited from the measurement of the above-mentioned judgment criteria during his pre- and post-operative consultations.

Exclusion Criteria:

* Presence in the medical file of the subject's opposition to the reuse of his data for scientific research purposes.
* Prolonged use of stored eye drops;
* Documented etiology of chronic alteration of the ocular surface (shingles, herpes, Gougerot-Sjogren syndrome, graft-versus-host disease);
* Minor patient or under guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years) operated on for cataract at HUS between January 2022 and January 2024;
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04-22 (Estimated)

PRIMARY OUTCOMES:
To assess whether cataract surgery induces an increased risk of corneal epithelial alterations in diabetic patients | One month before and one month after surgery
  The six Oxford scheme grades (0-5), which denote the severity of dry eye, are used to record the results:
  * Stage 0 or 1: Mild
  * Stage 2 or 3: Moderate
  * Stage 4 or 5: Severe

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Ophtalmologie - CHU de Strasbourg - France, Strasbourg, France

REFERENCES:
- [Derived] Koestel E, Dormegny L, Sauer A, Gaucher D, Bourcier T. Ocular surface changes and corneal epithelial remodeling after cataract surgery in patients with type 2 diabetes: a case-control study. BMC Ophthalmol. 2025 Jul 1;25(1):355. doi: 10.1186/s12886-025-04178-6. PMID 40597813